CLINICAL TRIAL: NCT03553446
Title: 50% Effective Concentration of Sevoflurane for Immobility in Cerebral Palsy Children Undergoing Botulinum Toxin Injection
Brief Title: 50% Effective Concentration of Sevoflurane for Immobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sung Mee Jung, Professor, Yeungnam University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YUMC-2018-04-023
Record Dates: First submitted 2018-05-08; First posted 2018-06-12 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Anesthetics, Inhalation
Keywords: Sevoflurane; Motion; Botulinum toxins; Cerebral palsy
MeSH Terms: conditions — Respiratory Aspiration; Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children receiving sevoflurane (Experimental): Children receiving pre-determined sevoflurane concentration using modified Dixon's up-and-down method
  Interventions: Drug: children receiving sevoflurane

INTERVENTIONS:
Drug: children receiving sevoflurane — Children receiving pre-determined sevoflurane concentration using modified Dixon's up-and-down method

SUMMARY:
Sevoflurane is as attractive inhalation agent fore deep sedation in children undergoing short invasive procedure because of lack of irritation to the respiratory tract, a pleasant odor and rapid clinical effect and recovery due to low blood gas partition coefficient.

The aim of this study is to determine the optimum inspired concentration of sevoflurane required for immobility during botulinum toxin injection in spontaneously breathing children with cerebral palsy.

DETAILED DESCRIPTION:
All anesthetics were administered by a single experienced anesthesiologist. Anesthetic induction was performed progressively with inhaled 1-8% sevoflurane, if the patient was cooperative, otherwise directly to the 8%, and subsequent maintenance 2% in oxygen at 5 L /min. A face mask was connected to a Mapleson C circuit for it. Patients breathed spontaneously, unaided, via a pediatric face mask. A failure was defined as the patient continued to move after following the study protocol for sevoflurane inhalation. Insufficient sedation was treated with increments of 0.5% concentration to achieve the desired effect, ie, maintenance of immobility during botulinum toxin injection. The sevoflurane concentration in the next patient would be adjusted depending on the success or failure for immobility at given sevoflurane concentration ( if successful, 0.5% lower concentration, if failed, 0.5% higher concentration).

The child was recovered from sevoflurane sedation at the end of botulinum toxin injection and transferred to post-anesthetic care unit.

ELIGIBILITY:
Inclusion Criteria:

* 3-12 years old children with cerebral palsy receiving sevoflurane inhalation for botulinum toxin injection
* American society of anesthesiologists Physical status 1-2

Exclusion Criteria:

* Body mass index > 30 kg/m2
* unstable heart disease
* Anticipated difficult airway history including congenital facial or airway anomaly
* Recent upper respiratory tract infection ( < 2 weeks)
* Gastroesophageal reflux
* Allergy history to sevoflurane, remifentanil or any drug used during procedure

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2018-07-29 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
the incidence of immobility | during procedure (Botulinum injection)
  cerebral palsy child who maintains immobility during botulinum toxin injection

CONTACTS AND LOCATIONS:
Overall Officials: Sung Mee Jung, M.D.,PhD., Principal Investigator — Yeungnam University Hospital
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

REFERENCES:
- [Derived] Kim K, Lee E, Jung SM, Baek J. 50% effective concentration of sevoflurane for immobility in cerebral palsy children undergoing botulinum toxin injection. Medicine (Baltimore). 2022 Oct 21;101(42):e30928. doi: 10.1097/MD.0000000000030928. PMID 36281165